CLINICAL TRIAL: NCT03430778
Title: Effect of Pneumoperitoneum on the Continuous and Non-invasive Hemoglobin Monitoring for Laparoscopic Gastrectomy: a Randomized Controlled Study
Brief Title: Effect of Pneumoperitoneum on the Continuous and Non-invasive Hemoglobin Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-17-339
Record Dates: First submitted 2018-02-01; First posted 2018-02-13 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High CO2 group (Experimental): end tidal CO2 : 40-45 mmHg
  Interventions: Other: High end-tidal CO2
- Low CO2 group (Placebo Comparator): end tidal CO2 : 30-35 mmHg
  Interventions: Other: Low CO2 group

INTERVENTIONS:
Other: High end-tidal CO2 — maintaining of end-tidal CO2 with the range of 40-45 mmHg
  Arms: High CO2 group
Other: Low CO2 group — maintaining of end-tidal CO2 with the range of 30-35 mmHg
  Arms: Low CO2 group

SUMMARY:
The primary purpose of this study is to investigate the effect of pneumoperitoneum on the continuous and non-invasive hemoglobin monitoring during laparoscopic gastrectomy

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic gastrectomy under general anesthesia

Exclusion Criteria:

* atypical hemoglobin disease, infective state, cardiovascular disease, peripheral vascular disease

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
difference between SpHb value and SaHb value (SpHb - SaHb) | from the start of anesthesia to the end of anesthesia, an average 2 hours
  SpHb value is measured by co-oxymetry, and SaHb value is measured by blood sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoum, South Korea